CLINICAL TRIAL: NCT04251949
Title: Evaluation of Photobiomodumation Using LED Lamp as a Curative Treatment for Oral or Oropharyngeal Mucositic Inducted by Radiation Therapy
Brief Title: Evaluation of the Photobiomodulation Using LED Lamp for Curative Treatment of Radio-induced Mucositis.
Acronym: MuciLight
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Oscar Lambret (Other)
Collaborators: Fondation Apicil (Other); Santelys Association (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MuciLight-1903; 2020-A00976-33 (Other: ANSM)
Record Dates: First submitted 2020-01-03; First posted 2020-02-05 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-12

CONDITIONS: Oral Cancer; Oropharyngeal Cancer
Keywords: Oral cancer; Radiotherapy; Radio-chemotherapy; Mucositis; LED photobiomodulation (PLED); Oropharyngeal cancer
MeSH Terms: conditions — Mouth Neoplasms; Oropharyngeal Neoplasms; Mucositis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: LED photobiomodulation — 1 PLED session before each radiotherapy session, until the end of the radio or radio-chemotherapy treatment. Each session will last 7 minutes. The light delivered will be preset on the lamp which will deliver a red light of a wavelength of 630nm, at a fluence of 37J/cm².

SUMMARY:
This is a monocentric, prospective, non-comparative phase II study with minimal risks and constraints. The study will aim to assess the curative treatment of radio-induced mucositis by photobiomodulation using LED lamp.

DETAILED DESCRIPTION:
The aim of this study is to assess the effectiveness of the treatment of radio- or radio-chemotherapy-induced early stage mucositis (stage 1 and 2) by photobiomodulation using LED lamp (PLED) in terms of controlling the mucositis assessed at the end of radiotherapy or radio-chemotherapy treatment.

Other objectives of the study include:

* To assess the pain evolution over-time, both overall over the evaluation period until the end of radiotherapy and at each session
* To assess the needs of level 3 analgesics (morphine, oxycodone, fentanyl, hydromorphone) during the PLED protocol.
* To assess the quality of life variation between inclusion and the end of treatment by radiotherapy or radio-chemotherapy.
* To estimate the frequency of radiotherapy or radio-chemotherapy treatment (temporary or permanent interruption, dose modification), and eventually, the reason of this modification.
* To assess the feasibility of photobiomodumation by LED (PLED) in this context.
* To assess the tolerability of photobiomodumation by LED (PLED) in a short term.
* To assess the frequency of the needs of nutritional support by nasogastric tube or gastrostomy tube during the PLED protocol.
* To assess the weight and general condition variation during the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* With squamous cell carcinoma of the head and/or neck
* Stage 1 or 2 mucositis (NCI-CTCAE v5), wich means a mucositis not requiring an enteral nutrition management (solid or liquid alimentation possible, including with feed supplements) in week 2 to 4 in relation to the beginning of radiotherapy.
* During treatment by radiotherapy, with or without concomitant chemotherapy
* Patient affiliated to a social security system
* Patient who signed the informed consent for this study

Exclusion Criteria:

* Radiotherapy treatment completed
* Stage 3 or higher mucositis already installed
* History of skin porphyria or lupus erythematosus
* Concomitant or within 7 days prior to inclusion, at least one of following drugs : fluoroquinolones, cycline, methotrexate, auranofine
* Enteral nutrition support in progress
* Pregnant or breast-feeding woman
* Patient under guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2021-03-19 (Actual); Primary Completion 2022-09-19 (Actual); Study Completion 2022-09-19 (Actual)

PRIMARY OUTCOMES:
Mucositis assessment | Change from baseline mucositis assessment at 7 weeks
  The mucositis will be assessed at least once a week between the inclusion and the end of treatment by radiotherapy or radio-chimiotherapy. It will be graded according to the NCI-CTCAE v5 scale. The scale ranging from 1 to 5. Where 1 is mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated and where 5 is death related to adverse event.
  We will consider as success the non-occurrence of stage 3 or higher mucositis between the inclusion and the end of radiotherapy. All patient presenting stage 3 or higher mucositis, which means, aphagia leading to an indication of nutritional support between the inclusion and the end of radiotherapy will be considered as a failure.
  A patient receiving less than 60 grey for an other reason than mucositis will be concidered as not assessable for the primery outcome.

SECONDARY OUTCOMES:
Pain related to the mucositis | At baseline, during each session - at least 3 times a week during 7 weeks, at the end of the study (week 7)
  Pain will be assessed with a decimal numerical scale (END) from 0 to 10. Where 0 is no pain felt and 10 is the maximal pain felt.
  An estimation of the average difference between each mesure will be performed.
Starting a level 3 analgesic treatment (morphine, oxycodone, fentanyl, hydromorphone) | Through study completion, an average of 7 weeks
  Percentage of patients starting a level 3 analgesic treatment during the study.
Quality of Life (QoL) | At baseline and at week 7 (end of the study)
  The quality of life will be evaluated using the EORTC-QLQ-C30 questionnaire. This questionnaire aim to assess the quality of life of cancer and it's composed of 30 questions.
  In this questionnaire, the items are scored from 1-4, where 1 = not at all, 2 = a little, 3 = quite a bit and 4 = very much.
  Only 2 items in the EORTC-QLQ-C30 questionnaire are scored from 1-7, where 1 is very poor and 7 is excellent.
  After that, questions from 31 to 65 are about H&N35, still to assess the quality of life of cancer.
  The items are scored from 1-4, where 1 = not at all, 2 = a little, 3 = quite a bit and 4 = very much.
  Only 5 items are scored from 1-2, where 1 = No and 2 = Yes.
Modification of treatment by radiotherapy or radio-chemotherapy | Through study completion, an average of 7 weeks
  Percentage of patient with an interruption (temporary or permanent) or dose modification.
Interruption of sessions | Through study completion, an average of 7 weeks
  Percentage of patient with session interruption, temporary or permanent.
Number of side effects | Through study completion, an average of 7 weeks
  Percentage of patients with side effect probably related to the photobiomodulation LED treatment.
Nutritional support by nasogastric tube or gastrostomy tube | Through study completion, an average of 7 weeks
  Percentage of patients with needs of nutritional support by nasogastric tube or gastrostomy tube.
Weight variation | Every week during the study (7 weeks)
  Weighting at each visit and comparison between the values
Performance status | Every week during the study (7 weeks)
  Assessment of the general condition by the scale of performance status (OMS) from 0 to 5.

CONTACTS AND LOCATIONS:
Overall Officials: Xavier XL LIEM, MD, Principal Investigator — Centre Oscar Lambret
Locations (1):
- Centre Oscar Lambret, Lille, France

IPD SHARING:
Plan to Share IPD: No